CLINICAL TRIAL: NCT04116112
Title: Blood Pressure After Endovascular Stroke Therapy-II: A Randomized Trial
Brief Title: Blood Pressure After Endovascular Stroke Therapy-II
Acronym: BEST-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Eva A. Mistry, Assistant Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 191520; K23NS113858 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-04 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Acute Stroke; Endovascular Thrombectomy
Keywords: Blood Pressure Control
MeSH Terms: conditions — Stroke | interventions — Nicardipine; Labetalol; Hydralazine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Higher Systolic Blood Pressure (SBP) Target (Experimental): Lower systolic blood pressure to ≤180 mmHg and maintain for 24 hours. If anti-hypertensive medication used, then maintain ≥160 mmHg.
  Interventions: Drug: Nicardipine; Drug: Labetalol; Drug: Hydralazine
- Lower SBP (<160 mmHg) Target (Experimental): Lower systolic blood pressure to <160 mmHg and maintain for 24 hours. If anti-hypertensive medication used, then maintain >140 mmHg.
  Interventions: Drug: Nicardipine; Drug: Labetalol; Drug: Hydralazine
- Lower SBP (<140mmHg) Target (Experimental): Lower systolic blood pressure to <140 mmHg and maintain for 24 hours. If anti-hypertensive medication used, then maintain >110 mmHg.
  Interventions: Drug: Nicardipine; Drug: Labetalol; Drug: Hydralazine

INTERVENTIONS:
Drug: Nicardipine — In the event where SBP values are above the randomly assigned target, intravenous nicardipine will be initiated at 2.5 mg/hr to lower the SBP. If SBP is still not reduced to below assigned target after 15 minutes, nicardipine dose will be increased by 2.5 mg/hr every 15 minutes until the target SBP or a maximum dose of 15 mg/hr is reached.
  Other Names: Cardene
Drug: Labetalol — If SBP is above target despite maximum nicardipine infusion for 30 minutes, 10-20 mg of intravenous labetalol will be added every 15 minutes.
Drug: Hydralazine — If SBP remains unresponsive for 1 hr despite the use of maximum doses of nicardipine and labetalol, a Hydralazine will be added at the treating physician's discretion. Incidence of the latter scenario is anticipated to be exceedingly rare.
  Other Names: Apresoline

SUMMARY:
The purpose of this study is to assess the safety of lowering blood pressure in acute stroke patients that are successfully treated with a mechanical thrombectomy procedure. The investogators will evaluate the hypothesis that lower blood pressure management strategies do not result in larger volume of stroke or worse 3-month clinical outcome in these patients.

DETAILED DESCRIPTION:
Several thousand patients suffer from an ischemic stroke caused by an occlusion of a large blood vessel supplying the brain. Endovascular mechanical thrombectomy (EVT) has revolutionized management of this most devastating type of ischemic stroke by allowing removal of the occlusive clot. However, about half of the successfully EVT-treated patients (~85% of all treated patients) still remain disabled at 90 days. Early evidence suggests that patients with lower blood pressure (BP) after the thrombectomy procedure have better outcomes. However, safety of lowering BP in these patients has not been determined. The primary safety concern of lowering BP comes from the potential of compromising blood flow to the "at risk" area of the brain following the stroke.

The purpose of this trial is to evaluate the safety of lower BP management strategies in patients who are successfully treated with endovascular treatment for ischemic stroke. The investigator will enroll 120 individuals who qualify and randomly assign them to one of the three systolic BP (SBP) targets: ≤180 mmHg, <160 mmHg, and <140 mmHg (40 patients in each group). Treatment will begin soon after the blood clot causing the stroke is removed, using anti-hypertensive medication given intravenously with a goal to lower and maintain the SBP below assigned target for 24 hrs.

The scientists will assess the safety of lower BP targets (<160 mmHg and <140 mmHg) by quantifying the volume of stroke measured with an MRI scan obtained at 36+/-12 hours and participants' functional status at 90 days measured with a patient centered disability score. Participants will undergo the 36 +/-12-hour MRI scan as part of their routine clinical care and will not be asked to prolong their hospital stay for study purpose. A phone interview will take place to determine their functional status at 90-days.

Enrollment of 120 patients will provide 80% power to detect a 10 cubic centimeter increase in stroke volume and a 0.10 decrease in utility-weighted modified Rankin score (a patient-centered disability score) for every 20 mmHg decrease in SBP. An interim analysis will be conducted after enrollment of 60 patients at which time the study may stop for safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Undergoing successful EVT (defined as modified Thrombolysis in Cerebral Ischemia Score, mTICI, ≥2b) for an occlusion in the anterior cerebral circulation large vessel (internal carotid artery and M1 or M2 segments of the middle cerebral artery).
* Intervention will be initiated only for those with a successful recanalization (modified Thrombolysis in Cerebral Ischemia Score ≥ 2b).
* Undergoing a baseline CT or MR perfusion study
* Those with unsuccessful recanalization (mTICI 0-2a) will be not intervened upon.

Exclusion Criteria:

* Known heart failure with ejection fraction <30%
* Presence of a left ventricular assist device
* Patients undergoing extracorporeal membrane oxygenation
* Pregnancy
* Enrollment in any other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Mistry, MBBS, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - Hartford Healthcare, Hartford, Connecticut
  - University of Cincinnati, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Mistry EA, Hart K, Davis T, Yeatts S, Lindsell CJ, Lewis RJ, Albers G, Wanderer JP, Prestigiacomo C, Bernard GR, Khatri P. Design of the BEST-II Randomized Clinical Trial. Stroke Vasc Interv Neurol. 2022 May 5;2(3):e000249. doi: 10.1161/SVIN.121.000249. eCollection 2022 May. PMID 41583626
- [Derived] Mistry EA, Hart KW, Davis LT, Gao Y, Prestigiacomo CJ, Mittal S, Mehta T, LaFever H, Harker P, Wilson-Perez HE, Beasley KA, Krothapalli N, Lippincott E, Stefek H, Froehler M, Chitale R, Fusco M, Grossman A, Shirani P, Smith M, Jaffa MN, Yeatts SD, Albers GW, Wanderer JP, Tolles J, Lindsell CJ, Lewis RJ, Bernard GR, Khatri P. Blood Pressure Management After Endovascular Therapy for Acute Ischemic Stroke: The BEST-II Randomized Clinical Trial. JAMA. 2023 Sep 5;330(9):821-831. doi: 10.1001/jama.2023.14330. PMID 37668620

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
Started | 40 | 40 | 40
Completed | 39 | 36 | 38
Not Completed | 1 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target | Total
Number analyzed (Participants) | 40 | 40 | 40 | 120
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [58 to 76.3] | 70.5 [61.8 to 76] | 74 [66.8 to 84.8] | 71 [62.8 to 77]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 20 | 21 | 28 | 69
  Male | 19 | 19 | 12 | 50
  Unknown | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Race | 5 | 2 | 2 | 9
  White Race | 34 | 37 | 34 | 105
  Multi-racial | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Other | 1 | 1 | 0 | 2
Alberta Stroke Program Early CT score [Median (Inter-Quartile Range); unit: Scores on a Scale] — ASPECT score is a score on a scale that ranges from 0 to 10. 0 denotes a larger stroke size and 10 denotes a smaller stroke size.
  Scores on a Scale | 8 [7 to 9] | 7 [6 to 8] | 8 [7 to 9] | 8 [7 to 9]
Pre-stroke modified Rankin score [Median (Inter-Quartile Range); unit: units on a scale, 0-6 (6=death)] | 0 [0 to 1] | 0 [0 to 0.25] | 0.5 [0 to 2] | 0 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Final Infarct Volume
Description: Infarct volume on diffusion-weighted MRI (or CT if MRI cannot be obtained) at 36 (+/-12) hrs after treatment initiation, adjusted for the baseline CT perfusion core infract volume.
Time Frame: 36 (+/-12) hrs after treatment initiation
Measure: Mean (95% Confidence Interval); unit: Cubic Centimeters
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
Number analyzed (Participants) | 39 | 36 | 38
Cubic Centimeters | 46.4 [24.5 to 68.2] | 50.7 [33.7 to 67.7] | 32.4 [18.0 to 46.7]

2. Primary Outcome: Utility-weighted Modified Rankin Score
Description: Modified Rankin score (mRS) is a scale for measuring the degree of disability or dependence of people who have suffered a stroke. 0 - no symptoms at all; 1 - no significant disability despite symptoms; able to carry out all usual duties and activities; 2- slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance; 3- moderate disability; requiring some help, but able to walk without assistance; 4 - moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance; 5 - severe disability; bedridden, incontinent and requiring constant nursing care and attention; 6- dead.
  Patient centered utility weights are applied to these scores as 1.0 for mRS level 0; 0.91 for mRS level 1; 0.76 for mRS level 2; 0.65 for mRS level 3; 0.33 for mRS level 4; 0 for mRS level 5; and 0 for mRS level 6. Unlike the mRS, the utility-weighted mRS runs from 0 to 1, with 0 being the worst.
Time Frame: 90 days after treatment initiation
Measure: Mean (95% Confidence Interval); unit: units on a scale (Range 0-1; 1=best)
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
Number analyzed (Participants) | 37 | 39 | 37
units on a scale (Range 0-1; 1=best) | 0.58 [0.46 to 0.71] | 0.47 [0.35 to 0.6] | 0.51 [0.38 to 0.63]

3. Secondary Outcome: Number of Participants With Any Hemorrhagic Transformation
Description: Number of participants with any new bleeding within the infarcted brain tissue on 36(+/-12) hr MRI/CT scan after treatment initiation
Time Frame: 36(+/-12) hrs after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
Number analyzed (Participants) | 40 | 37 | 39
Participants | 12 | 12 | 14

4. Secondary Outcome: Number of Participants With Symptomatic Hemorrhagic Transformation
Description: Defined as number of participants with any new bleeding within the infarcted brain tissue and an NIH Stroke Scale worsening of 4 or more points associated with the bleeding within 36 (+/-12) hrs of treatment initiation
Time Frame: 36(+/-12) hrs after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
Number analyzed (Participants) | 37 | 35 | 37
Participants | 2 | 1 | 2

5. Secondary Outcome: Number of Participants With Neurological Worsening Associated With Antihypertensive Treatment
Description: Defined as number of participants with 4 points of greater increase in NIH Stroke scale associated with reduction in SBP caused by anti-hypertensive treatment initiation or titration.
Time Frame: Treatment initiation to 24 hrs after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
Number analyzed (Participants) | 40 | 40 | 40
Participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Compliance Outcome
Description: Number of participants with an hourly maximum SBP above target from 2-24 hrs post treatment initiation
Time Frame: Treatment initiation to 24 hrs after treatment Initiation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through hospital stay, up to 30 days
Arm/Group | Higher Systolic Blood Pressure (SBP) Target | Lower SBP (<160 mmHg) Target | Lower SBP (<140mmHg) Target
All-Cause Mortality (participants affected / at risk) | 3/40 | 6/40 | 3/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 3/40 | 4/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Systolic Blood Pressure (SBP) Target (N=40) | Lower SBP (<160 mmHg) Target (N=40) | Lower SBP (<140mmHg) Target (N=40)
Femoral artery Pseudoaneurysm (Vascular disorders) | 1 | 0 | 0
Sepsis and cardiac failure (Infections and infestations) | 0 | 1 | 0
Aspiration Pneumonia (Infections and infestations) | 0 | 2 | 0
Carotid artery re-occlusion (Vascular disorders) | 0 | 0 | 1
Subarachnoid hemorrhage (Nervous system disorders) | 0 | 0 | 1
Gastrointestinal hemorrhage associated with gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
New contralateral large vessel occlusion stroke (Nervous system disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Participants enrolled at only three sites across the US

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT04116112/Prot_SAP_000.pdf